CLINICAL TRIAL: NCT01315119
Title: The Role of SPY Intra-Operative Angiography in Determining Adequate Skin Perfusion in Immediate Breast Reconstruction With Implants
Brief Title: SPY Intra-Operative Angiography & Skin Perfusion in Immediate Breast Reconstruction w/ Implants
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BRS0005; BRS0005 (Other: Stanford University)
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: SPY Intra-Operative Angiography — Calculated per patient
  Other Names: Novadaq SPY

SUMMARY:
The investigators hope to learn the value of the SPY ELITE® intra-operative angiography in reducing post-operative complications associated with low breast skin blood flow after breast reconstruction using implants.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women, and over 180,000 women will be diagnosed with this disease in 2008. Last year, over 57,000 breast reconstructive procedures were performed, of which prosthetic reconstruction constituted 76%. Immediate reconstruction has been favored over delayed procedures for psychological and technical reasons. However, immediate breast reconstruction is associated with significantly higher complication rates (50-52%) than delayed procedures (32-36%), especially when a prosthetic technique is used. For prosthetic reconstructions, the most significant early complications include necrosis of the mastectomy skin flaps, infection, delayed wound healing and exposure of the implant. The published incidence of these complications ranges between 10% and 40% and is predominantly associated with malperfusion of mastectomy skin flaps. Thus, evaluation of skin perfusion and elimination of poorly vascularized areas could help reduce the high rate of complications in immediate breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

3.1.0 Ability to understand and the willingness to sign a written informed consent document.

3.1.1 Signed written informed consent.

3.1.2 Women with local or regional recurrences after previous breast conserving surgery.

3.1.3 Women undergoing delayed post mastectomy reconstruction.

3.1.4 Women undergoing prophylactic mastectomy.

3.1.5 Women with invasive or non-invasive breast cancer, receiving breast conserving surgery with or without reduction mammoplasty or mastectomy, with or without immediate reconstruction.

3.1.6 Women of 18 years of age or older.

3.1.7 ECOG or Karnofsky Performance Status 0,1,2.

3.1.8 Basic Metabolic Panel within 6 months

3.1.9 Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Exclusion Criteria:

3.2.1 History of liver or kidney failure will not be eligible.

3.2.2 Allergies to iodine containing products will not be eligible.

3.2.3 Women who are pregnant will not be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population includes women with unilateral or bilateral breast cancer undergoing immediate or delayed breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09-23 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | During surgery
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | Immediately post operative
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | 2 weeks
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | 1 month
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | 3 months
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | 6 months
To compare clinical visual assessment of skin viability with intraoperative SPY imaging. | 12 months

SECONDARY OUTCOMES:
Establish the percentage of patients with ischemia or necrosis in the first year post surgery. | 12 months
Number and type of complications in the first year. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C. Gurtner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States